CLINICAL TRIAL: NCT07014345
Title: Double-Lumen Tube Intubation in the Lateral Position Versus the Supine Position on First-Attempt Success Rate Among Patients Undergoing Thoracic Surgery: A Prospective, Randomized, Controlled, Multi-center Trial
Brief Title: Double-Lumen Tube Intubation in the Lateral Position Versus the Supine Position on First-Attempt Success Rate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar studies have been conducted
Sponsor: xiangming fang (Other)
Collaborators: Red Cross Hospital, Hangzhou, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Central People's Hospital of Zhanjiang (Other); The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor-Investigator, xiangming fang, Chair Professor, Department of Anesthesiology Vice Dean, School of Medicine and and Pharmaceutical sciences Zhejiang University, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intubation
Record Dates: First submitted 2025-05-22; First posted 2025-06-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Double Lumen Tube Intubation
Keywords: Double-lumen tube; lateral position intubation; first-attempt success rate; thoracic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DLT placement performed in lateral position (Experimental): In the lateral position group, patients were positioned laterally (as required for surgery) before anesthesia induction. After anesthesia induction, Double lumen tube placement was performed while the patient remained in the lateral position.
  Interventions: Procedure: DLT placement performed in lateral position
- DLT placement performed in supine position (No Intervention): A double-lumen tube is typically carried out with the patient in the supine position, which is a standard procedure in thoracic surgery.

INTERVENTIONS:
Procedure: DLT placement performed in lateral position — In the lateral position group, patients were positioned laterally (as required for surgery) before anesthesia induction. After anesthesia induction, Double lumen tube placement was performed while the patient remained in the lateral position.
  Arms: DLT placement performed in lateral position

SUMMARY:
The aim of this clinical trial is to find out the first success rate of double lumen intubation in the lateral position in thoracic surgery, it will also find out the safety of double lumen tube intubation in the lateral position. The trial aims to answer the following key questions

Does intubation in lateral position improve the first-time success rate of double-lumen intubation compared with in the supine position? What medical problems can participants experience during double lumen tube intubation in the lateral position? The researchers will compare double lumen intubation in the lateral position vs supine position to see if the position is effective in the success rate of double lumen intubation.

Participants will

Use the supine or lateral position during intubation

ELIGIBILITY:
Inclusion Criteria:

* need for DLT intubation with elective unilateral thoracoscopic surgery
* age 18-65 years
* American Society of Anesthesiologists (ASA) grade of I or II
* no serious cardiopulmonary disease

Exclusion Criteria:

* aged <18 years or >65 years
* body mass index >30 kg/m2
* cognitive dysfunction and inability to assume the required body position
* previous cervical vertebrae and expected difficult airway (e.g., Mallampati airway grade of III, IV, or higher, maximum mouth opening <3 finger widths, nail-chin distance <6 cm)
* admission to the intensive care unit after surgery and without follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Successful First-Pass Intubation | Periprocedural
  The primary outcome was the success rate of the first DLT intubation attempt.

SECONDARY OUTCOMES:
No. of intubation attempts | Periprocedural
  Number of patients who were successfully intubated on any attempt
Intubation time | Periprocedural
  Defined as from the time when the laryngoscope passed between the patient's lips until the use of a fiberoptic bronchoscope to confirm the correct positioning of the DLT.
Interval before surgery | Periprocedural
  Defined as the time interval between the admission of patients in the operating room and the start of surgery.
p-Peak | Periprocedural
  peak inspiratory pressure(p-Peak) during mask ventilation, total-lung ventilation(TLV) and one-lung ventilation(OLV)
Flexible bronchoscope usage | Periprocedural
  the frequency of use of flexible bronchoscope
the incidence of DLT malposition | Periprocedural
  the incidence of DLT malposition observed by flexible bronchoscope (DLT malposition was defined as movement >1.0 cm to correct the DLT position)
early intubation-related complications | Periprocedural
  early intubation-related complications (dental injury; hypoxemia; laryngospasm; bronchospasm; airway trauma; arrhythmia, including the salve of ventricular premature beats, ventricular fibrillation, and ventricular tachycardia; oral mucosal injury; and esophageal intubation)
postoperative complications | Periprocedural
  postoperative complications (sore throat, GRBAS scale, upper-arm discomfort, and nerve injury)
satisfaction scores. | Periprocedural
  0 points: dissatisfied, 1 point: satisfied, 2 points: very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Kim H, Seol T, Han SH, Kim H, Hwang JY. A bench study on the prevention of lung-to-lung aspiration with double-lumen endobronchial tubes and bronchial blockers. Sci Rep. 2024 Jan 2;14(1):187. doi: 10.1038/s41598-023-50792-z. PMID 38167877
- [Background] Campos JH. Lung isolation techniques for patients with difficult airway. Curr Opin Anaesthesiol. 2010 Feb;23(1):12-7. doi: 10.1097/ACO.0b013e328331e8a7. PMID 19752725
- [Background] Brodsky JB. Lung separation and the difficult airway. Br J Anaesth. 2009 Dec;103 Suppl 1:i66-75. doi: 10.1093/bja/aep262. PMID 20007992
- [Background] Yang M, Kim JA, Ahn HJ, Choi JW, Kim DK, Cho EA. Double-lumen tube tracheal intubation using a rigid video-stylet: a randomized controlled comparison with the Macintosh laryngoscope. Br J Anaesth. 2013 Dec;111(6):990-5. doi: 10.1093/bja/aet281. Epub 2013 Aug 23. PMID 23975566
- [Background] Saji H, Okada M, Tsuboi M, Nakajima R, Suzuki K, Aokage K, Aoki T, Okami J, Yoshino I, Ito H, Okumura N, Yamaguchi M, Ikeda N, Wakabayashi M, Nakamura K, Fukuda H, Nakamura S, Mitsudomi T, Watanabe SI, Asamura H; West Japan Oncology Group and Japan Clinical Oncology Group. Segmentectomy versus lobectomy in small-sized peripheral non-small-cell lung cancer (JCOG0802/WJOG4607L): a multicentre, open-label, phase 3, randomised, controlled, non-inferiority trial. Lancet. 2022 Apr 23;399(10335):1607-1617. doi: 10.1016/S0140-6736(21)02333-3. PMID 35461558